CLINICAL TRIAL: NCT03120403
Title: Safety and Efficacy of Intrathecal Morphine in Children Undergoing Major Abdominal Surgeries, Dose-finding Clinical Study
Brief Title: Safety and Efficacy of Intrathecal Morphine in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alaa Ali Mohamed Elzohry (Other)
Responsible Party: Sponsor-Investigator, Alaa Ali Mohamed Elzohry, Lecturer in South Egypt Cancer Insitute, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: intrathecal morphine
Record Dates: First submitted 2017-04-10; First posted 2017-04-19 (Actual); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Abdominal Cancer

STUDY DESIGN:
Intervention Model Description: intratehcal injection of drug( morphine).
Who Masked: Participant, Investigator
Masking Description: using opaque sealed envelopes containing computer generated randomization schedule, the opaque sealed envelopes are sequentially numbered that were open before application of anesthetic plan.
Oversight: US Export: Yes

ARMS (3):
- intrathecal morphine 2 μg/kg (Active Comparator): After G A and securing the tube in place , the patients will be placed in the lateral decubtious position and a single dose of intrathecal morphine will be performed using a 25 gauge needle (Brown ®,Germany) and free flow of CSF technique.children will receive intrathecal morphine 2 μg/kg in 2 ml volume normal saline.
  Interventions: Procedure: intrathecal morphine
- intrathecal morphine 5 μg/kg (Active Comparator): After G A and securing the tube in place , the patients will be placed in the lateral decubtious position and a single dose of intrathecal morphine will be performed using a 25 gauge needle (Brown ®,Germany) and free flow of CSF technique. children will receive intrathecal morphine 5 μg/kg in 2 ml volume normal saline.
  Interventions: Procedure: intrathecal morphine
- intrathecal morphine 10 μg/kg (Active Comparator): After G A and securing the tube in place , the patients will be placed in the lateral decubtious position and a single dose of intrathecal morphine will be performed using a 25 gauge needle (Brown ®,Germany) and free flow of CSF technique.children will receive intrathecal morphine 10 μg/kg in 2 ml volume normal saline.
  Interventions: Procedure: intrathecal morphine

INTERVENTIONS:
Procedure: intrathecal morphine

SUMMARY:
Postoperative pain in pediatrics can usually be well controlled with a combination of analgesics including acetaminophen ( paracetamol) ,NSIADS, opioids , and local/regional anesthesia.The use of epidural and subarachnoid morphine for analgesia in adults has grown almost as quickly as Morton's discovery of anesthesia in 1846. The application of these techniques to the pediatric patients has evolved much more slowly,although significant progress is being made by many investigators.

DETAILED DESCRIPTION:
Advantage of intrathecal morphine as that extremely small doses of opioids are required when administrated intrathecally because they have direct access to spinal cord opioid receptors. Drug administered epidurally or caudally are required in much higher doses because they must first diffuse into the CSF before they reach spinal opioid receptors. As a result, the duration of action of intrathecal morphine is greater than that of single shot peridural techniques.

To investigate the safety and efficacy of intrathecal morphine in post operative pain relief in pediatric patients undergoing major abdominal cancer surgeries using different doses of intrathecal morphine (2 μg/kg , 5 μg/kg ,10μg/kg).

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients aged 3-12 years , weighting between 10-30 kg , and of American Society of Anesthesiologists (ASA) physical status I and II scheduled for major abdominal surgeries , expected to last more than 90 minutes under general anesthesia combined with intratehcal morphine.

Exclusion Criteria:

* Children with sacral bone abnormalities ,spina bifida , coagulopathy , mental delay or retardation , known allergy to the study drugs , and local infection at the site of injection will be excluded from the study.

Ages: 3 Years to 12 Years | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-03-30 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
The face , Legs , Activity, Crying , and Consolability (FLACC) score | 24 hours (every 4 hours )
  The face , Legs , Activity, Crying , and Consolability (FLACC) pain score with its 0- 10 score range will be used to assess pain

IPD SHARING:
Plan to Share IPD: Undecided